CLINICAL TRIAL: NCT04358094
Title: Analgesia Assessment of Conversational Hypnosis Script During Peripherical Veinous Catheter Set up Versus Standard Script in Operating Room
Brief Title: Conversational Hypnosis for Peripherical Veinous Access (HYPNACESS)
Acronym: HYPNACESS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 2020-A00187-32
Record Dates: First submitted 2020-04-16; First posted 2020-04-22 (Actual); Last update posted 2020-04-22 (Actual); Status verified 2020-04

CONDITIONS: Vascular Access Site Pain

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conversational hypnosis script (Experimental): Patient who received conversational hypnosis script during peripherical veinous access set up
  Interventions: Other: Conversational hypnosis script
- Standard script (Other): Patient who received standard script during peripherical veinous access set up
  Interventions: Other: Standard script

INTERVENTIONS:
Other: Conversational hypnosis script — Conversational hypnosis during peripherical veinous catheter set up
  Arms: Conversational hypnosis script
Other: Standard script — Standard script during peripherical veinous catheter set up
  Arms: Standard script

SUMMARY:
The peripherical veinous catheterization is required for anesthesia. However, it's a painful procedure and causes stress or even phobia.

Hypnosis can be seen as an interesting tool. Conversational hypnosis needs no training. It is used by script, which makes it easier.

The working hypothesis for study is that the conversational hypnosia script reduces pain during the set up of peripherical veinous access.

The main objective is the analgesia assessment of conversational hypnosis script for peripherical veinous catheter set up versus standard script in operating room. A nurse anesthetist is reading the conversational script or standard script during the procedure. The nurse anesthetist is untrained for hypnosis.

The secondary objective are the level of anxiety, patient satisfaction within the perioperative period (EVAN G questionnaire), the heart rate and the evaluation how nurse anesthetist feels about using the script after each use.

ELIGIBILITY:
Inclusion Criteria:

* Digestive endoscopy procedure under general anesthesia in one of the participating centers
* Patient speaking and understanding French
* Patient affiliated or entitled to a social security scheme
* Patient who received enlightened information about the study and who co-signed, with the investigator, a consent to participate after a minimum period of reflection

Exclusion Criteria:

* Patient with deafness
* Patient with cognitive impairment
* Pregnant and / or breastfeeding patient
* Patient with dissociative disorders (contraindication to hypnosis)
* Patient suffering from a pathology which can cause chronic pain
* Patient receiving analgesia or anxiety drug
* Patient under justice, curatorship or tutorship
* Patient deprived of liberty by judicial or administrative decision

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 200 (Estimated)
Dates: Start 2020-05-04 (Estimated); Primary Completion 2020-12-30 (Estimated); Study Completion 2021-01-18 (Estimated)

PRIMARY OUTCOMES:
Analgesia assessment by digital pain scale | immediately after applying the peripherical veinous catheter dressing
  Digital pain scale: it describes the severity of the pain On this scale, "0" represents "no pain" and "10" represents "the worst possible pain"

SECONDARY OUTCOMES:
Level of anxiety by numerical scale | before randomization and immediately after peripherical veinous catheter set up
  Digital scale: it describes the severity of the pain On this scale, "0" represents "no anxiety" and "10" represents "the worst possible anxiety"
patient satisfaction within the perioperative period (EVAN G questionnaire) | between 4 and 48 hours after the procedure
  EVAN G questionnaire: Score from 0 to 100
  The higher the score, the higher the level of patient satisfaction
Heart rate | during the procedure
  maximum heart rate
Nurse anesthetist feeling about using the script after each use by digital scale | immediately after procedure
  Evaluate how nurse anesthetist feels about using the script after each use by digital scale ranging from 0 to 10.
  On this scale, "0" represents " uncomfortable" and "10" represents " very comfortable "

CONTACTS AND LOCATIONS:
Overall Officials: Hervé Bouaziz, Pr, Principal Investigator — Central Hospital, Nancy, France
Locations (1):
- Centre Hospitalier Régional Universitaire, Nancy, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Armstrong P, Young C, McKeown D. Ethyl chloride and venepuncture pain: a comparison with intradermal lidocaine. Can J Anaesth. 1990 Sep;37(6):656-8. doi: 10.1007/BF03006485. PMID 2208537
- [Background] Nir Y, Paz A, Sabo E, Potasman I. Fear of injections in young adults: prevalence and associations. Am J Trop Med Hyg. 2003 Mar;68(3):341-4. PMID 12685642
- [Background] Ferreira-Valente MA, Pais-Ribeiro JL, Jensen MP. Validity of four pain intensity rating scales. Pain. 2011 Oct;152(10):2399-2404. doi: 10.1016/j.pain.2011.07.005. PMID 21856077
- [Background] Auquier P, Pernoud N, Bruder N, Simeoni MC, Auffray JP, Colavolpe C, Francois G, Gouin F, Manelli JC, Martin C, Sapin C, Blache JL. Development and validation of a perioperative satisfaction questionnaire. Anesthesiology. 2005 Jun;102(6):1116-23. doi: 10.1097/00000542-200506000-00010. PMID 15915023